CLINICAL TRIAL: NCT06181045
Title: A Phase 1, Single-Ascending-Dose, Randomized, Double-Blind Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3410738 in Healthy Adult Subjects
Brief Title: A Study of LY3410738 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LOXO-IDH-20003; I9Y-OX-JDHD (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Treatment A): LY3410738 (Experimental): Single oral dose of LY3410738 or placebo administered as over-encapsulated capsule formulation.
  Interventions: Drug: LY3410738; Drug: Placebo
- Cohort 2 (Treatment B): LY3410738 (Placebo Comparator): Single oral dose of LY3410738 or placebo administered as over-encapsulated capsule formulation.
  Interventions: Drug: LY3410738; Drug: Placebo
- Cohort 3 (Treatment C): LY3410738 (Experimental): Single oral dose of LY3410738 or placebo administered as over-encapsulated capsule or tablet formulation.
  Interventions: Drug: LY3410738; Drug: Placebo
- Cohort 4 (Treatment D): LY3410738 (Experimental): Single oral dose of LY3410738 or placebo administered as over-encapsulated capsule or tablet formulation.
  Interventions: Drug: LY3410738; Drug: Placebo
- Cohort 5 (Treatment E): LY3410738 (Experimental): Single oral dose of LY3410738 or placebo administered as over-encapsulated capsule or tablet formulation.
  Interventions: Drug: LY3410738; Drug: Placebo
- Cohort 6 (Treatment F): LY3410738 (Experimental): Single oral dose of LY3410738 or placebo administered as over-encapsulated capsule or tablet formulation.
  Interventions: Drug: LY3410738; Drug: Placebo
- Cohort 7 (Treatment G): LY3410738 (Experimental): Single oral dose of LY3410738 or placebo administered as over-encapsulated capsule or tablet formulation.
  Interventions: Drug: LY3410738; Drug: Placebo

INTERVENTIONS:
Drug: LY3410738 — Administered orally.
Drug: Placebo — Administered orally.

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of LY3410738 and to look at the amount of the study drug, LY3410738, that gets into the blood stream and how long it takes the body to get rid of it when given in healthy adult participants. For each participant, the total duration of the study will be 53 days, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive
* Male and female participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods
* Must comply with all study procedures, including the 3-night stay at the Clinical Research Unit (CRU) and follow-up phone call

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Positive serologic test for hepatitis B surface antigen (HBsAg), hepatitis B virus immunoglobulin M (HBV IgM) core antibody, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening.
* Positive polymerase chain reaction (PCR) test for COVID-19 at Screening
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee)
* Have previously received LY3410738 in any other study investigating LY3410738, within 30 days prior to Day 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through 53 days
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to 24 Hours Post-dose (AUC0-24) of LY3410738 | Pre-dose up to 24 hours post-dose
  PK: AUC0-24 of LY3410738
PK: Area Under the Concentration-time Curve, From Time 0 to the Last Measurable Concentration (AUC0-t) of LY3410738 | Pre-dose up to 48 hours post-dose
  PK: AUC0-t of LY3410738
PK: Maximum Observed Plasma Concentration (Cmax) of LY3410738 | Pre-dose up to 48 hours post-dose
  PK: Cmax of LY3410738
PK: Time to Maximum Observed Plasma Concentration (Tmax) of LY3410738 | Pre-dose up to 48 hours post-dose
  PK: Tmax of LY3410738

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo-Avrutin, Study Director — Loxo Oncology, Inc.
Locations (2):
- United States (2):
  - Covance Clinical Research Unit, Daytona Beach, Florida
  - Covance Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No